CLINICAL TRIAL: NCT07076797
Title: The Effects of Lower Extremity Functional Exercise Program and Neuromuscular Electrical Nerve Stimulation on Muscle Strength, Muscle Thickness, Gait and Fall Risk in the Elderly
Brief Title: Effects of Lower Extremity Functional Exercise Program and Neuromuscular Electrical Nerve Stimulation in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Ugur Cavlak, PROF. PhD, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BiruniUniversityIst
Record Dates: First submitted 2025-07-01; First posted 2025-07-22 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Neuromuscular Electrical Stimulation
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: a randomized controlled study.
Who Masked: Participant
Masking Description: The participants will not know the group distrubution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1-NMES (Experimental): experimental group will receive neuromuscular electrical stimulation
  Interventions: Other: NMES
- Group 2-EXERCISE (Active Comparator): acticve comparator group will receive exercise training
  Interventions: Other: EXERCISE TRAINING

INTERVENTIONS:
Other: EXERCISE TRAINING — PHYSIOTHERAPY PROGRAM
  Arms: Group 2-EXERCISE
Other: NMES — PHYSIOTHERAPY PROGRAM
  Arms: Group 1-NMES

SUMMARY:
The aim of this study was to investigate and compare the effects of lower extremity functional exercise program and neuromuscular electrical nerve stimulation on muscle thickness, muscle strength, gait and fall risk in the elderly.

DETAILED DESCRIPTION:
Study Design: It will be a randomized, controlled study. The participants to be included in the study will be divided into two groups using the random randomization method. In this method; participants will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Relatively healthy older women aged 65-84 years
* Individuals without neurological, orthopedic, systemic (cardiovascular) problems that would prevent them from performing the test
* To have a score of 6 and above on the Hodkinson Abbreviated Mental Test
* At least 90 points on the Barthel activities of daily living test
* Ability to walk independently (with or without walking aids)
* Living in a nursing home or in their own home

Exclusion Criteria:

* Having a defined neurological (including vertigo), orthopedic, orthopedic, psychiatric, systemic (cardiovascular, cachectic due to malnutrition) disease that prevents walking and mobility
* Being in the statin drug group
* Diagnosis of sarcopenia
* Having communication problems
* Visual impairment (severe) or hearing impairment (severe)

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Imaging | baseline and week 13
  Thickness measurements for both lower extremity quadriceps femoris muscle and tibialis anterior muscle will be evaluated. For resting muscle thickness, the person will be positioned in a supine position with the knee extended and the leg in neutral rotation (weights will be placed on the ankles to prevent external rotation laterally). The distance between the spina iliaca anterior superior and the upper border of the patella on the anterior thigh region will be measured with a tape measure, the probe will be placed transversely on the long axis of the thigh so that it is 1/3 of the distance close to the patella, and this area will be marked with a pencil. When evaluating the tibialis anterior muscle, the patient will be in the supine position at a point corresponding to 30% of the distance between the lateral tibial condyle and the lateral malleolus. Transmission gel will be used between the skin and the ultrasound head.
Assessment of Muscle Strength | bbaseline and week 13
  Quadriceps and tibialis anterior muscle strength will be measured with digital handheld dynamometer. The digital muscle measurement device is a portable device with 3 interchangeable heads and a digital LCD screen. The device can provide data such as Peak power, time to reach peak power, total test time and average force in kg Newton and pounds. For the measurement of Quadriceps strength on both legs; the test will begin with the participants sitting on a flat surface with their hips and knees flexed at 90 degrees. The dynamometer will be placed perpendicular to the leg, 1-2 cm above the level of the malleoli. The "make test" technique, which requires isometric contraction, will be applied. All measurements will be taken twice from both legs of the participants by the same researcher with the same hand. For the Tibialis anterior strength measurement on both legs, the participant will be asked to dorsiflex their ankles while lying face down on a flat table.

SECONDARY OUTCOMES:
10-Meter Walking Test | baseline and week 13
  During the test, the patient will walk at a normal walking speed between two markers that are 10 meters apart and the elapsed time will be recorded. Measurements will be made twice and the best value will be recorded. The number of steps in a 10-meter distance during walking will also be recorded (Wade, 1992)
Dynamic Balance Test (Timed Up and Go Test) | baseline and week 13
  The timed up and go test will be used. The test evaluates functional mobility, balance and performance in older adults. The patient, wearing normal shoes and conventional walking aids, begins the test in a standard chair with his back leaning, his arms resting on the arms of the chair and both feet flat on the floor. The patient is asked to stand up and walk to a line on the floor 3 meters away, turn on the line, walk back to the chair and sit on the chair (Shumway, 2000). The test ends when the patient's hip touches the chair. The test is repeated twice; the fastest time is recorded. <10 s of movement, >13.5 s means an increased risk of falling (Podsiadlo, 1991; Şahin, 2008).
Static Balance Test (One-Legged Standing Test) | baseline and week 13
  One-Legged Standing Test The one-legged standing test (eyes open) will be used. One leg is lifted without touching the standing leg. The eyes remain open and the patient is asked to maintain their balance for 30 seconds (Stevenson, 1996). If the lifted leg touches the supporting leg, if the lifted leg touches the ground, the patient is asked to.
Sit-to-Stand Chair Test | baseline and week 13
  İt will also be used to evaluate lower extremity muscle strength. The patient sits on a chair without arm support, the patient tries to do 5 sit-stands with a signal the person is allowed 2 attemps and the fastes score is recorded.
Assessment of Fall Risk | baseline and week 13
  The Fullerton Balance Scale (FAB-T) will be used. It was developed to identify more subtle changes in multiple dimensions of balance.
Participant Satisfaction Assessment | baseline and week 13
  a satisfaction assessment consisting of 0-10 points will be made for both groups before and after the intervention for elderly individuals. The two extreme definitons of the parameter to be evaluated 0 and 10 points. The patients written on both ends of a 100 mm line and will be asked to indicate where his/her situation is appropriate on this line by drawing a line putting a dut or pointing.

CONTACTS AND LOCATIONS:
Overall Officials: UGUR CAVLAK, Prof., Principal Investigator — Biruni University
Locations (1):
- Faculty of Health Sciences in Biruni University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cadore EL, Casas-Herrero A, Zambom-Ferraresi F, Idoate F, Millor N, Gomez M, Rodriguez-Manas L, Izquierdo M. Multicomponent exercises including muscle power training enhance muscle mass, power output, and functional outcomes in institutionalized frail nonagenarians. Age (Dordr). 2014 Apr;36(2):773-85. doi: 10.1007/s11357-013-9586-z. Epub 2013 Sep 13. PMID 24030238
- [Background] Sarabon N, Kozinc Z, Lofler S, Hofer C. Resistance Exercise, Electrical Muscle Stimulation, and Whole-Body Vibration in Older Adults: Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Clin Med. 2020 Sep 8;9(9):2902. doi: 10.3390/jcm9092902. PMID 32911822

DOCUMENTS (2):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Study protocol (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT07076797/Prot_SAP_ICF_000.pdf
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: PROTOCOL and ICF (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT07076797/Prot_SAP_ICF_001.pdf